CLINICAL TRIAL: NCT01016873
Title: A Double-masked, Sham Controlled, Dose-ranging Study to Evaluate the Safety and Effectiveness of Low Voltage Stereotactic Radiosurgery in Patients With Choroidal Neovascularization (CNV) Secondary to Age-related Macular Degeneration (AMD)
Brief Title: INTREPID - IRay Plus Anti-VEGF Treatment For Patients With Wet AMD
Acronym: INTREPID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oraya Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLH002
Record Dates: First submitted 2009-11-19; First posted 2009-11-20 (Estimated); Results first posted 2014-12-05 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: AMD; Wet AMD; Age-Related Macular Degeneration; Wet Age-Related Macular Degeneration; Macular Degeneration; Eye Diseases; Retinal Diseases
Keywords: Oraya; Oraya Therapeutics, Inc.; low voltage stereotactic radiotherapy; radiotherapy; IRay; Ranibizumab; Lucentis; AMD; Macular Degeneration; xray; radiation; x ray; external beam radiation; radiosurgery
MeSH Terms: conditions — Macular Degeneration; Eye Diseases; Retinal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 16 Gy IRay (Experimental): 16 Gy IRay + PRN Lucentis®
  Interventions: Device: IRay
- Sham 16 Gy IRay (Sham Comparator): Sham 16 Gy IRay + PRN Lucentis®
  Interventions: Device: IRay
- 24 Gy IRay (Experimental): 24 Gy IRay + PRN Lucentis®
  Interventions: Device: IRay
- Sham 24 Gy IRay (Sham Comparator): Sham 24 Gy IRay + PRN Lucentis®
  Interventions: Device: IRay

INTERVENTIONS:
Device: IRay — Low voltage stereotactic radiotherapy system

SUMMARY:
The purpose of this study is to confirm the safety and establish the effectiveness of two doses from the IRay System for the treatment of wet AMD.

DETAILED DESCRIPTION:
The purpose of this study is to confirm the safety of low voltage external beam radiotherapy using the IRay System at two dose levels for the treatment of CNV secondary to neovascular AMD and to determine if the IRay System is effective in sparing the number of Lucentis injections during the first 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have neovascular AMD diagnosed within the previous 3 years, have received at least 3 injections with Lucentis® or Avastin® within the previous year and have the need for treatment with anti-VEGF therapy due to increased fluid or persistent cysts on OCT, or leakage on FA.
* Patients must have a total lesion size of <12 disc areas and a CNV lesion with the greatest linear dimension of <6 mm, but not greater than 3 mm from the center of the fovea to the furthest point on the lesion perimeter.
* The distance from the center of the fovea to the nearest edge of the optic disc should be not less than 3 mm.
* Patients must Patient must be at least 50 years of age.
* Women must be post-menopausal ≥1 year or surgically sterilized, or a pregnancy screen must be performed prior to the study and a reliable form of contraception approved by the investigator must be maintained during the study.
* Patient must have best corrected visual acuity of 75 to 25 letters in the study eye and at least 20 letters in the fellow eye.

Exclusion Criteria:

* CNV due to causes other than AMD, including ocular histoplasmosis syndrome, angioid streaks, multifocal choroiditis, choroidal rupture, or pathologic myopia (spherical equivalent ≥ -8 diopters).
* An axial length of ≤20 mm or ≥26 mm.
* Previously diagnosed with Diabetes Mellitus and/or an HbA1c of >6.5%, and with retinal findings consistent with diabetic retinopathy.
* Prior or concurrent therapies for age related macular degeneration including submacular surgery, subfoveal thermal laser photocoagulation (with or without photographic evidence), transpupillary thermotherapy (TTT), ocular photodynamic therapy, radiation therapy to the head or neck in the study eye.
* Previous posterior vitrectomy, or any surgery in the study eye within 6 months or YAG capsulotomy within 3 months prior to the screening visit.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2009-11; Primary Completion 2012-05 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denis O'Shaughnessy, Ph.D., Study Director — Oraya Therapeutics, Inc.
Locations (21):
- Austria (4):
  - LKH Graz, Graz
  - Universitätsklinik Innsbruck, Innsbruck
  - Hanusch Krankenhaus Wien, Vienna
  - Ordination Prof. Michael Stur, Vienna
- Czechia (6):
  - Fakultni Nemocnice Brno, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni Nemocnice Olomouc, Olomouc
  - Faculty Hospital Kralovske Vinohrady, Prague
  - General Faculty Hospital Prague, Prague
  - Military Hospital Prague, Prague
- Germany (3):
  - Kopfklinikum University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg
  - University Eye Hospital, Tübingen, Baden-Wurttemberg
  - Klinik für Augenheilkunde, Neubrandenburg, Mecklenburg-Vorpommern
- Università Vita-Salute Istituto Scientifico San Raffaele, Milan, Italy
- United Kingdom (7):
  - Royal Victoria Hospital, Belfast
  - Bradford Royal Infirmary, Bradford
  - Torbay Hospital, Devon
  - King's College, London
  - Manchester Royal Eye Hospital, Manchester
  - Southampton General Hospital, Southampton
  - Royal Wolverhampton Hospital NHS Foundation Trust, Wolverhampton

REFERENCES:
- [Derived] Evans JR, Igwe C, Jackson TL, Chong V. Radiotherapy for neovascular age-related macular degeneration. Cochrane Database Syst Rev. 2020 Aug 26;8(8):CD004004. doi: 10.1002/14651858.CD004004.pub4. PMID 32844399

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham IRay: Sham 24 or 16 Gy IRay + PRN Lucentis®
  IRay: Low voltage stereotactic radiotherapy system
Period: 12 Months
Arm/Group | 16 Gy IRay | 24 Gy IRay | Sham IRay
Started | 75 | 75 | 80
Completed | 74 | 72 | 79
Not Completed | 1 | 3 | 1
Period: 24 Months
Arm/Group | 16 Gy IRay | 24 Gy IRay | Sham IRay
Started | 74 | 72 | 79
Completed | 69 | 68 | 73
Not Completed | 5 | 4 | 6
Period: 36 Months
Arm/Group | 16 Gy IRay | 24 Gy IRay | Sham IRay
Started | 69 | 68 | 73
Completed | 58 | 64 | 67
Not Completed | 11 | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Sham IRay: Sham 16 or 24 Gy IRay + PRN Lucentis®
  IRay: Low voltage stereotactic radiotherapy system
- Total: Total of all reporting groups
Arm/Group | 16 Gy IRay | 24 Gy IRay | Sham IRay | Total
Number analyzed (Participants) | 75 | 75 | 80 | 230
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 73.35 (7.18) | 73.77 (8.26) | 73.45 (7.14) | 73.52 (7.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 48 | 49 | 140
  Male | 32 | 27 | 31 | 90
Region of Enrollment [Number; unit: participants]
  Czech Republic | 48 | 29 | 47 | 124
  Austria | 4 | 20 | 4 | 28
  Germany | 6 | 7 | 10 | 23
  United Kingdom | 14 | 18 | 17 | 49
  Italy | 3 | 1 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Lucentis® Injections Up To And Including Week 52
Time Frame: During the first 52 weeks.
Measure: Mean (Standard Deviation); unit: Injections
Arm/Group | 16 Gy IRay | 24 Gy IRay | Sham IRay
Number analyzed (Participants) | 75 | 75 | 80
Injections | 2.64 (2.46) | 2.44 (2.41) | 3.73 (2.58)

2. Secondary Outcome: Change in Mean Visual Acuity (VA)
Time Frame: Weeks 12, 28, 52 and 104.
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | 16 Gy IRay | 24 Gy IRay | Sham IRay
Number analyzed (Participants) | 75 | 75 | 80
Letters
  Visual Acuity (VA) - Baseline | 57.91 (12.72) | 58.75 (12.79) | 59.29 (13.09)
  Mean change in VA Week 12, n = 73, 71, 78 | 0.86 (5.68) | 1.85 (9.73) | 2.06 (6.79)
  Mean change in VA Week 28, n = 73, 73, 77 | -0.33 (8.25) | 2.04 (8.58) | 1.42 (7.91)
  Mean change in VA Week 52, n = 74, 72, 79 | -0.28 (8.77) | 0.40 (10.33) | -0.58 (10.56)
  Mean change in VA Week 104, n = 68, 68, 73 | -10.03 (16.45) | -7.49 (16.49) | -6.71 (17.08)

3. Secondary Outcome: Percentage (Pct.) of Patients (Pts.) Losing < 15 Letters of Best Correct Visual Acuity (BCVA) From Baseline (Base.)
Time Frame: Weeks 12, 28 and 52.
Population: Number of Participants Analyzed:
  * Week 12: n = 73, 71, 78
  * Week 28: n = 73, 73, 77
  * Week 52: n = 74, 72, 79
Measure: Number; unit: Percentage of Patients
Arm/Group | 16 Gy IRay | 24 Gy IRay | Sham IRay
Number analyzed (Participants) | 75 | 75 | 80
Percentage of Patients
  Pct. of Pts. Losing <15 Letters From Base. - W12 | 100 | 97 | 97
  Pct. of Pts. Losing <15 Letters From Base. - W28 | 97 | 96 | 97
  Pct. of Pts. Losing <15 Letters From Base. - W52 | 93 | 89 | 92

4. Secondary Outcome: Percentage (Pct.) of Patients (Pts.) Gaining ≥ 15 Letters of Best Correct Visual Acuity (BCVA) From Baseline (Base.)
Time Frame: Weeks 12, 28 and 52.
Population: Number of Participants Analyzed:
  * Week 12: n = 73, 71, 78
  * Week 28: n = 73, 73, 77
  * Week 52: n = 74, 72, 79
Measure: Number; unit: Proportion of Patients
Arm/Group | 16 Gy IRay | 24 Gy IRay | Sham IRay
Number analyzed (Participants) | 75 | 75 | 80
Proportion of Patients
  Pct. of Pts. Gaining >=15 Letters from Base. -W12 | 0 | 6 | 1
  Pct. of Pts. Gaining >=15 Letters from Base. -W28 | 4 | 4 | 3
  Pct. of Pts. Gaining >=15 Letters from Base. -W52 | 4 | 4 | 5

5. Secondary Outcome: Percentage (Pct.) of Patients (Pts.) Gaining ≥ 0 Letters of Best Correct Visual Acuity (BCVA) From Baseline (Base.)
Time Frame: Weeks 12, 28 and 52.
Population: Number of Participants Analyzed:
  * Week 12: n = 73, 71, 78
  * Week 28: n = 73, 73, 77
  * Week 52: n = 74, 72, 79
Measure: Number; unit: Percentage of Patients
Arm/Group | 16 Gy IRay | 24 Gy IRay | Sham IRay
Number analyzed (Participants) | 75 | 75 | 80
Percentage of Patients
  Pct. of Pts. Gaining >=0 Letters From Base. - W12 | 60 | 65 | 74
  Pct. of Pts. Gaining >=0 Letters From Base. - W28 | 52 | 62 | 64
  Pct. of Pts. Gaining >=0 Letters From Base. - W52 | 53 | 57 | 57

6. Secondary Outcome: Time From Mandatory Injection at Day 0 to the First PRN Injection.
Time Frame: 52 Weeks
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | 16 Gy IRay | 24 Gy IRay | Sham IRay
Number analyzed (Participants) | 75 | 75 | 80
Weeks | 16.29 [12.14 to 20.29] | 16.71 [12.57 to 26.29] | 13.14 [12.14 to 16.14]

7. Secondary Outcome: Total Number (No.) of Lucentis® Injections (Inject.) During The First 12, 28, and 104 Weeks.
Time Frame: Week 12, 28, and 104
Measure: Mean (Standard Deviation); unit: Number of Injections
Arm/Group | 16 Gy IRay | 24 Gy IRay | Sham IRay
Number analyzed (Participants) | 75 | 75 | 80
Number of Injections
  Mean No. of Injections - Week 12, n = 75,75,80 | 0.57 (0.70) | 0.56 (0.74) | 0.73 (0.78)
  No. of Injections - Week 28, n = 75,75,80 | 1.51 (1.35) | 1.28 (1.37) | 1.83 (1.41)
  Mean No. of Injections - Week 104, n=75,75,80 | 4.48 (3.94) | 5.37 (4.57) | 6.61 (4.28)

8. Secondary Outcome: Mean Change in Choroidal Neovascularization (CNV) as % of Lesion on Fluorescein Angiography (FA) From Baseline to Week 52
Time Frame: Week 52
Measure: Mean (Standard Deviation); unit: CNV as % of Lesion
Arm/Group | 16 Gy IRay | 24 Gy IRay | Sham IRay
Number analyzed (Participants) | 29 | 28 | 44
CNV as % of Lesion | -0.16 (0.33) | -0.18 (0.33) | -0.10 (0.26)

ADVERSE EVENTS:
Time Frame: Adverse event reporting from Baseline through week 104.
Arm/Group | 16 Gy IRay | 24 Gy IRay | Sham IRay
Serious Adverse Events (participants affected / at risk) | 12/75 | 8/75 | 7/80
Other Adverse Events (participants affected / at risk) | 20/75 | 23/75 | 24/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 16 Gy IRay (N=75) | 24 Gy IRay (N=75) | Sham IRay (N=80)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Choroidal neovascularisation (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal Vein Occlusion (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Intracranial haematoma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary bladder polyp (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Colpocele (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Limb operation (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0)
Cyst drainage (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Foot operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 16 Gy IRay (N=75) | 24 Gy IRay (N=75) | Sham IRay (N=80)
Worsening of macular degeneration (Eye disorders) | 7 (7) | 6 (6) | 8 (8)
Retinal haemorrhage (Eye disorders) | 4 (4) | 2 (2) | 6 (6)
Visual acuity reduced (Eye disorders) | 5 (5) | 3 (3) | 4 (4)
Blepharitis (Eye disorders) | 2 (2) | 7 (7) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 7 (7) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and the Principal Investigator agree not to publish or issue a press release or authorize the publication or presentation of any Study Results without obtaining Oraya's prior written approval.